CLINICAL TRIAL: NCT07266337
Title: Clinical Study on the Safety and Efficacy of CD19/BCMA CAR T-cell Therapy for Refractory Systemic Lupus Erythematosus
Brief Title: CD19/BCMA CAR-T for SLE
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chengdu Ucello Biotechnology Co., Ltd. (Industry)
Collaborators: The General Hospital of Western Theater Command (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCAR-SLE
Record Dates: First submitted 2025-11-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: SLE - Systemic Lupus Erythematosus
Keywords: SLE; CAR-T
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells treatment (Experimental)
  Interventions: Drug: CD19/BCMA CAR T-cells

INTERVENTIONS:
Drug: CD19/BCMA CAR T-cells — intravenous injection of CD19/BCMA CAR-T cells

SUMMARY:
The purpose of this clinical trial is to learn if CD19/BCMA CAR-T works to treat refractory SLE in adults. It will also learn about the safety and efficacy of the CD19/BCMA CAR-T cell product.

The main questions it aims to answer are:

1. What CAR-T-related adverse events (AEs) occur within 3 months after the CAR-T cell infusion?
2. Which dose level is the optimal biological dose (OBD)?
3. What is the the changes of disease activity status, proportion of patients achieving DORIS remission, percentage of participants achieving maintenance of drug-free DORIS remission, proportion of patients achieving SRI-4 remission, percentage of participants achieving maintenance of LLDAS?

Participants will:

1. Receive CD19/BCMA CAR-T cells infusion on Day 0.
2. Be hospitalized for at least 7 days post-infusion for close safety monitoring and remain within 2 hours of the treatment facility for at least 28 days.
3. Visit the clinic at Day 14, Day 28, month 3, month 6, month 9, month 12, month 18 and month 24 after CAR-T cells infusion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years (inclusive), regardless of gender.
* Definitive diagnosis of systemic lupus erythematosus (SLE) meeting the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for SLE
* Treatment refractory: failed ≥ 2 Conventional SLE treatments for at least 3 months.
* Disease activity assessed by SELENA-SLEDAI score ≥ 6 with at least one British Isles Lupus Assessment Group (BILAG)-2004 Class A (severe manifestation) or two Class B (moderate manifestation) organ scores (or both); OR SELENA-SLEDAI score ≥ 8.
* Adequate function of major organs as follows:

Bone marrow function: a. Neutrophil count ≥ 1×10⁹/L (no colony-stimulating factor therapy within 2 weeks prior to testing, excluding neutropenia caused by SLE); b. Hemoglobin ≥ 60 g/L.

Liver function: Alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN) (excluding ALT elevation caused by SLE); Aspartate aminotransferase (AST) ≤ 3 × ULN (excluding AST elevation caused by SLE); Total bilirubin (TBIL) ≤ 1.5 × ULN (excluding TBIL elevation caused by SLE).

Renal function: Creatinine clearance rate (CrCl) ≥ 30 mL/minute (calculated by Cockcroft/Gault formula, excluding CrCl reduction caused by SLE).

Coagulation function: International normalized ratio (INR) ≤ 1.5 × ULN; Prothrombin time (PT) ≤ 1.5 × ULN.

Cardiac function: Hemodynamically stable.

* Female subjects of childbearing potential and male subjects whose partners are of childbearing potential must use medically approved contraceptive methods or abstain from sexual intercourse during the study treatment period and for at least 6 months after the end of study treatment. Female subjects of childbearing potential must have a negative serum human chorionic gonadotropin (HCG) test within 7 days prior to study enrollment and must not be breastfeeding.
* Voluntarily agrees to participate in the clinical study, signs the informed consent form (ICF), and demonstrates good compliance with study procedures and follow-up.

Exclusion Criteria:

* History of severe drug allergies or atopic diathesis.
* Presence or suspicion of uncontrolled or treatment-requiring fungal, bacterial, viral, or other infections.
* Cardiac function insufficient to tolerate the study treatment.
* Congenital immunoglobulin deficiency.
* History of malignant tumors within the past 5 years.
* End-stage renal failure.
* Positive for hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA titer above the lower limit of detection; positive for hepatitis C virus (HCV) antibody with positive peripheral blood HCV RNA; positive for human immunodeficiency virus (HIV) antibody; positive syphilis test.
* History of mental illness or severe cognitive impairment.
* Use of disease-modifying immunosuppressive agents within 5 half-lives or biological agents within 4 weeks prior to enrollment.
* Pregnant females or females planning to become pregnant.
* Other conditions deemed by the investigator to preclude study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence rate of Dose limited toxicity (DLTs) | Up to 28 days after CD19/BCMA CAR-T injection
the incidence rate of CAR-T-related adverse events | up to 28 days after CD19/BCMA CAR-T injection

SECONDARY OUTCOMES:
Systemic Lupus Erythematosus Disease Activity Index score | month 6, month 9, month 12, month18, month 24 post CAR-T injection
  SLEDAI score
Proportion of patients achieving DORIS remission | month 6, month 9, month 12, month18, month 24 post CAR-T injection
Percentage of participants achieving maintenance of drug-free DORIS remission | month 6, month 9, month 12, month18, month 24 post CAR-T injection
Proportion of patients achieving SRI-4 remission | month 6, month 9, month 12, month18, month 24 post CAR-T injection
Percentage of participants achieving maintenance of LLDAS | month 6, month 9, month 12, month18, month 24 post CAR-T injection
British Isles Lupus Assessment Group 2004 score | month 6, month 9, month 12, month18, month 24 post CAR-T injection
  BILAG2004 score
Physician's Global Assessment score | month 6, month 9, month 12, month18, month 24 post CAR-T injection
  PGA score

OTHER OUTCOMES:
AUC of CAR-T cells | up to 2 months after CAR-T injection
  AUC is defined as the area under the curve in 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, M.D., Principal Investigator — The General Hospital of Western Theater Command
Locations (1):
- The General Hospital of Western Theater Command, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
The safety and efficacy data will be shared in a publication.